CLINICAL TRIAL: NCT02501720
Title: Comparison of Outcome of Post Burn Flexion Contracture Release Under Tourniquet Verses Tumescent Technique in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Muhammad Mustehsan Bashir, Associate professor of Plastic Surgery, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2335
Record Dates: First submitted 2015-07-12; First posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Hand Burns; Flexion Contracture
Keywords: burn; hand; flexion contracture; tourniquet; tumescent technique; children
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tourniquet Group (Active Comparator): Post burn flexion contractures will be released under tourniquet control
  Interventions: Procedure: post burn flexion contractures release under tourniquet control; Procedure: Contracture release and application of FTSG
- Tumescent technique group (Experimental): Post burn flexion contractures will be released using Tumescent solution
  Interventions: Procedure: post burn flexion contractures release using tumescent solution; Procedure: Contracture release and application of FTSG

INTERVENTIONS:
Procedure: post burn flexion contractures release under tourniquet control — post burn flexion contractures will be released under tourniquet control
  Arms: Tourniquet Group
Procedure: post burn flexion contractures release using tumescent solution — post burn flexion contractures will be released using tumescent solution
  Arms: Tumescent technique group
Procedure: Contracture release and application of FTSG — Post burn flexion contractures will be released and full thickness skin graft(FTSG) will be applied.

SUMMARY:
Post burn flexion contractures are common in pediatric age group. Release of contracture and coverage with full thickness skin graft (FTSG) is a widely used procedure for this problem. This procedure is routinely done under tourniquet control because bloodless operative field is essential to visualize important neurovascular structures in hand.

Use of tumescent technique without a tourniquet is gaining acceptance because it avoids complications associated with tourniquet use, maintains a blood less surgical field and decreases operative time. Furthermore use of tumescent anesthesia often results in better surgical outcomes.

Although the benefits of tumescent technique used in wide awake hand surgery are well documented, epinephrine at a concentration of 1:1 000,00 has also been used as a replacement for pneumatic tourniquet for release of hand contracture in infants and adults under general anesthesia. Thus epinephrine 1:1,000,00 in saline solution can be a potential replacement for a tourniquet in hand surgeries done under general anesthesia.

DETAILED DESCRIPTION:
Post burn flexion contractures are common in pediatric age group. Release of contracture and coverage with full thickness skin graft (FTSG) is a widely used procedure for this problem. This procedure is routinely done under tourniquet control because bloodless operative field is essential to visualize important neurovascular structures in hand.

Use of tumescent technique without a tourniquet is gaining acceptance because it avoids complications associated with tourniquet use, maintains a blood less surgical field and decreases operative time. Furthermore use of tumescent anesthesia often results in better surgical outcomes.

Although the benefits of tumescent technique used in wide awake hand surgery are well documented, epinephrine at a concentration of 1:1 000,000 has also been used as a replacement for pneumatic tourniquet for release of hand contracture in infants and adults under general anesthesia. Thus epinephrine 1:1,000,000 in saline solution can be a potential replacement for a tourniquet in hand surgeries done under general anesthesia.

To the investigators' knowledge no study has so far been done to compare the outcome of release of post burn flexion contractures under tumescent technique with general anesthesia or under tourniquet control with general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Children with post burn flexion contractures involving volar aspect of palm and fingers
* Possible to cover the defect with full thickness skin graft
* age range of 3 to 12 years.
* Patients of both genders

Exclusion Criteria:

* Children with recurrent post burn contractures.
* Children with any history of bleeding diathesis or coagulopathy.
* Children with any co-morbid condition making any contraindication of general anesthesia.
* Patients having previous history of vascular insufficiency like Raynaud's disease or phenomenon, severe peripheral vascular disease and peripheral neuropathy.
* The patient having allergic hypersensitivity to epinephrine, lidocaine.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Operative time to secure graft | Time of surgery
  Operative time to secure graft will be measured by calculating the time taken to secure per square centimeter of graft.
  Time (T) in minutes to secure per cm2 of graft = Total operative time / size of graft secured in cm2 measured by transparent graft paper In tourniquet group total operative time will be measured as total time taken from start of applying tourniquet including time taken for exsanguinations to the time till completion of dressing.
  In tumescent group total operative time will be measured as total time taken from start of injecting the tumescent solution including waiting time for tumescent solution to produce maximum vasoconstriction (25 minutes) to the time till completion of dressing
Percentage graft taken | 14th day post surgery
  It will be measured by the percentage of graft take at 14th post-operative day. Percentage graft take = Graft secured at the time of operation measured by using transparent graph paper / graft take at 14th post-operative day measured by using transparent graph paper.
Post-operative pain (FLACC scale) | At First hour after arrival in ward following surgery
  Post-operative pain will be measured by blinded on duty doctor using Face Leg Activity Cry Consolability (FLACC) scale. Postoperative pain will be measured by using FLACC pain scale by blinded observer at first hour postoperatively taking time of arrival in the ward as zero hour
Post-operative pain (FLACC scale) | At 6th hour after arrival in ward following surgery
  Post-operative pain will be measured by blinded on duty doctor using Face Leg Activity Cry Consolability (FLACC) scale. Postoperative pain will be measured by using FLACC pain scale by blinded observer at 6th hour postoperatively taking time of arrival in the ward as zero hour.
Post-operative pain (FLACC scale) | At 12th hour after arrival in ward following surgery
  Post-operative pain will be measured by blinded on duty doctor using Face Leg Activity Cry Consolability (FLACC) scale. Postoperative pain will be measured by using FLACC pain scale by blinded observer at 12th hour postoperatively taking time of arrival in the ward as zero hour.
Post-operative pain (FLACC scale) | At 24th hour after arrival in ward following surgery
  Post-operative pain will be measured by blinded on duty doctor using Face Leg Activity Cry Consolability (FLACC) scale. Postoperative pain will be measured by using FLACC pain scale by blinded observer at 24th hour postoperatively taking time of arrival in the ward as zero hour.

REFERENCES:
- [Background] Spuy L. Complications of arterial tourniquet. South Afr J Anaesth Analg. 2012; 18: 14-18.
- [Background] Lalonde D, Martin A. Tumescent local anesthesia for hand surgery: improved results, cost effectiveness, and wide-awake patient satisfaction. Arch Plast Surg. 2014 Jul;41(4):312-6. doi: 10.5999/aps.2014.41.4.312. Epub 2014 Jul 15. PMID 25075350
- [Background] Lalonde D. Minimally invasive anesthesia in wide awake hand surgery. Hand Clin. 2014 Feb;30(1):1-6. doi: 10.1016/j.hcl.2013.08.015. Epub 2013 Nov 9. PMID 24286736
- [Background] Teo I, Lam W, Muthayya P, Steele K, Alexander S, Miller G. Patients' perspective of wide-awake hand surgery--100 consecutive cases. J Hand Surg Eur Vol. 2013 Nov;38(9):992-9. doi: 10.1177/1753193412475241. Epub 2013 Jan 24. PMID 23348603
- [Background] Al Youha S, Lalonde DH. Update/Review: changing of use of local anesthesia in the hand. Plast Reconstr Surg Glob Open. 2014 Jun 6;2(5):e150. doi: 10.1097/GOX.0000000000000095. eCollection 2014 May. PMID 25289343
- [Background] Prasetyono TO. Tourniquet-Free Hand Surgery Using the One-per-Mil Tumescent Technique. Arch Plast Surg. 2013 Mar;40(2):129-33. doi: 10.5999/aps.2013.40.2.129. Epub 2013 Mar 11. PMID 23533019
- [Background] Shridharani S, Manson P, Magarakis M et al. The safety and efficacy of epinephrine in hand surgery: a systematic review of the literature and international survey. European Journal of Plastic Surgery. 2014; 37: 183-188.
- [Background] Gumus N. Tumescent infiltration of lidocaine and adrenaline for burn surgery. Ann Burns Fire Disasters. 2011 Sep 30;24(3):144-8. PMID 22396674